CLINICAL TRIAL: NCT05680363
Title: Prospective Sibling Oocyte Study of a New Method to Improve Embryo Development in IVF/ICSI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fecundis S.A. (Other)
Responsible Party: Sponsor
Organization: Fecundis Lab SL (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fecundis_2
Record Dates: First submitted 2022-12-06; First posted 2023-01-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Sperm Preparation (Active Comparator): Sperm samples in the control group will undergo traditional processing in the lab prior to insemination.
  Interventions: Device: Standard Sperm Preparation
- HyperSperm (Experimental): Sperm samples in the experimental group will undergo product-specific processing in the lab prior to insemination.
  Interventions: Device: HyperSperm

INTERVENTIONS:
Device: HyperSperm — Multi-step sperm preparation
  Arms: HyperSperm
Device: Standard Sperm Preparation — Standard sperm preparation
  Arms: Standard Sperm Preparation

SUMMARY:
Prospective, multi-centric, split-sample, sibling oocyte study evaluating the safety and efficacy of a new method to prepare sperm samples for IVF (in vitro fertilization) / ICSI (intracytoplasmic sperm injection) compared to standard procedures.

ELIGIBILITY:
Female:

Inclusion Criteria:

* With ovarian reserve of between 8 and 30 antral follicles counting both ovaries
* Treatment planned for embryo transfer at the blastocyst stage

Exclusion Criteria:

* Any diagnosed sexually transmitted infection (STI)
* Diabetes or other metabolic disorders.
* Recurrent pregnancy loss (defined as >2 clinical pregnancies without live birth).
* Previous failures in two or more IVF cycles

Male:

Inclusion Criteria for IVF:

* Age: 20-55 years
* Fresh sample (not cryopreserved )
* Sperm motility (TOTAL) ≥ 40% in spermogram
* Normal sperm morphology (Kruger criteria) ≥ 4% in spermogram
* Sperm count after swim up ≥ 5x10^6
* Treatment planned for embryo transfer at the blastocyst stage

Inclusion Criteria for ICSI:

* Age: 20-55 years
* Fresh sample (not cryopreserved )
* Sperm concentration ≥ 10x10^6 /ml in spermogram
* Sperm motility (TOTAL) ≥ 20% in spermogram
* Normal sperm morphology (Kruger criteria) ≥ 3% in spermogram
* Treatment planned for embryo transfer at the blastocyst stage

Exclusion Criteria:

* Any diagnosed sexually transmitted infection (STI)
* Total failure of in vitro fertilization in previous cycles.

Ages: 20 Years to 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Development rate to blastocysts | Days 5-6 post insemination
  Total blastocysts / total fertilized oocytes

SECONDARY OUTCOMES:
Fertilization rate | Day 1 post insemination
  Total fertilized oocytes (formation of two pronuclei) / total inseminated oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Buffone, PhD, Principal Investigator — Fecundis Lab SL
Locations (4):
- Argentina (4):
  - In Vitro Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Pregna, Buenos Aires, Buenos Aires F.D.
  - WeFIV, Buenos Aires, Buenos Aires F.D.
  - Fertya, Rosario, Santa Fe Province

IPD SHARING:
Plan to Share IPD: No